CLINICAL TRIAL: NCT05476315
Title: Is Emergency Surgery Back to Pre-covid-19 Era? Our Cohort Study
Brief Title: Emergency Surgery During Covid Compared to Emergency Surgery During Pre-covid Period
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical Doctor, University of Foggia
Other Study IDs: 6
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Emergencies; Surgery; COVID-19
MeSH Terms: conditions — Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Emergency surgery during covid-19 pandemic — Patients undergoing emergency surgery during the covid period and compared with emergency interventions before the pandemic

SUMMARY:
The aim of this study is to analyze the trend of hospitalizations and how emergency operations have qualitatively and quantitatively changed in our Department of Medical and Surgical Sciences of the Foggia Hospital from 2019 (pre-covid era) to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent emergency surgery from March 2019 to May 2022

Exclusion Criteria:

* Patients underwent elective surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our cohort-study was conducted by analyzing four groups of patients admitted to the Department of Medical and Surgical Sciences of the Hospital of Foggia, Apulia southern part of Italy :
  * group 1: people admitted during the no-covid period from March 09th, 2019 to May 09th, 2019;
  * group 2: people admitted from March 09th, 2020 to May 09th, 2020;
  * group 3: people admitted from March 09th, 2021 to May 09th, 2021
  * group 4: people admitted from March 09th, 2022 to May 09th, 2022
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Is emergency surgery back to pre-covid-19 era? | From March 2019 to May 2022
  How emergency surgery has changed during covid pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Pavone, Principal Investigator — University of Foggia
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-07-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT05476315/Prot_000.pdf